CLINICAL TRIAL: NCT06922565
Title: Efficacy of Acupuncture in the Treatment of Moderate-to-severe Atopic Dermatitis: a Multicentre Randomised Sham-controlled Clinical Trial
Brief Title: Efficacy of Acupuncture in the Treatment of Moderate-to-severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20250403
Record Dates: First submitted 2025-03-31; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- acupuncture group (Experimental)
  Interventions: Device: acupuncture
- sham acupuncture group (Sham Comparator)
  Interventions: Device: sham acupuncture
- Alternate control group (No Intervention)

INTERVENTIONS:
Device: acupuncture — Subjects in the acupuncture group received traditional acupuncture. The needles were inserted to induce a sense of 'getting qi' and left in place for 30 minutes.
  Arms: acupuncture group
Device: sham acupuncture — Sterile disposable retractable needles and a fake placebo acupuncture device are used for sham acupuncture. The acupuncturist attached the base of the sham acupuncture device to the acupoints, and then inserted sterile disposable blunt-tipped retractable needles into the tubes; when the blunt tips touched the skin, the needles retracted into the handles, and there was no sensation of getting qi.
  Arms: sham acupuncture group

SUMMARY:
This study used a multicentre parallel three-armed randomised sham-controlled clinical trial methodology in order to objectively and normatively assess the efficacy of acupuncture on Quchi the Sea of Blood the Foot Sanli and the Sanyinjiao in the treatment of moderate-to-severe atopic dermatitis so as to obtain high-level evidence-based medical evidence.

This study adopts a multi-centre, parallel, three-armed, randomized, sham-controlled clinical trial method, and will be conducted at Yueyang Hospital of Integrative Medicine affiliated with Shanghai University of Traditional Chinese Medicine, Huashan Hospital affiliated with Fudan University, and Seventh People's Hospital affiliated with Shanghai University of Traditional Chinese Medicine. Eligible patients with moderate-to-severe AD will be divided into three groups using stratified block randomisation in the ratio of 2:2:1: the acupuncture group, the sham-acupuncture group and the waitlisted control group. The total observation period is 9 weeks, including a 1-week introduction period, a 4-week treatment period and a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for moderate to severe atopic dermatitis;

  * Age ≥18 and ≤75 years old gender is not limited; ③ Peak Pruritus Numerical Rating Scale (PP-NRS) score ≥4; ④ Voluntarily participate in this trial and sign the informed consent form.

Exclusion Criteria:

* Patients who are in the acute onset of the disease and have erosions exudates and secondary infections;

  * Patients who have participated in other clinical studies in the past 3 months or are participating in other clinical studies; ③ Patients with severe haematological diseases (e.g. platelet count <50×109 /L) and other serious diseases that may affect operation and efficacy;

    * Current systematic use of glucocorticosteroids discontinued for less than 7 days; immunosuppressants (cyclosporine methotrexate tretinoin etc.) discontinued for less than 1 month; dulprevirizumab discontinued for less than 1 month JAK inhibitors discontinued for less than 2 weeks;

      * Women who are pregnant or breastfeeding; ⑥ Patients with a history of acupuncture treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-03 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
SCORing atopic dermatitis（SCORAD） | This indicator will be measured at baseline day 1 (V2), day 27 ± 1 (V9), and day 56 ± 3 (V10).
  SCORAD range of 0 ~ 103 points.The condition is classified as mild, moderate or severe according to the score, with the higher the score, the more severe the condition.

SECONDARY OUTCOMES:
Patient Oriented Eczema Measure (POEM) | This indicator will be measured at baseline day 1 (V2), day 27 ± 1 (V9), and day 56 ± 3 (V10).
  Patients themselves assessed the frequency and severity of 7 symptoms occurring in the past 1 week, with each entry on a 5-point scale corresponding to a score of 0, 1, 2, 3, and 4. Scores ranged from 0 ~ 28, with higher scores indicating greater severity.
Dermatology Life Quality Index（DLQI） | This indicator will be measured at baseline day 1 (V2), day 27 ± 1 (V9), and day 56 ± 3 (V10).
  The questionnaire contains 10 questions. Scores range from 0 to 30, with higher scores indicating a greater impact on quality of life.
Peak Pruritus Numerical Rating Scale（PP-NRS） | This indicator will be measured at baseline day 1 (V2), day 27 ± 1 (V9), and day 56 ± 3 (V10).
  The PP-NRS is a patient self-report, with a score of 0 for no itching and 10 for the worst itching imaginable, with the patient scoring the worst itching experienced in the last 24 h. The PP-NRS is a patient self-report, with a score of 0 for no itching and 10 for the worst itching imaginable.
Skin Peripheral sympathetic nerve activity (SKNA) | This indicator will be measured at baseline day 1 (V2), day 27 ± 1 (V9).
  Measured with neuECG, SKNA in µV
Serum total IgE | This indicator will be measured at baseline day 1 (V2), day 27 ± 1 (V9).
Peripheral blood serum cytokines（IL-4,IL-13,IL-31,IL-33,INF-α） | This indicator will be measured at baseline day 1 (V2), day 27 ± 1 (V9).